CLINICAL TRIAL: NCT00358566
Title: "Primovax" - A Phase III Trial Comparing GV1001 and Gemcitabine in Sequential Combination to Gemcitabine Monotherapy in Advanced Un-Resectable Pancreatic Cancer.
Brief Title: GV1001 and Gemcitabine in Sequential Combination to Gemcitabine Monotherapy in Pancreatic Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Preliminary data showed no survival benefit in the GV1001 group compared to the gemcitabine group.
Sponsor: Pharmexa A/S (Industry)
Collaborators: ICON Clinical Research (Industry); ORION Clinical Services (Industry); CIRION Central Laboratory (Unknown); Dorevitch (Unknown); Syneos Health (Other)
Responsible Party: Ask Aabenhus, Clinical Trial Manager, Pharmexa A/S
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PX115.1.1-302; Eudract no. 2005-005014-21
Expanded Access: Available
Record Dates: First submitted 2006-07-14; First posted 2006-08-01 (Estimated); Last update posted 2008-05-19 (Estimated); Status verified 2008-05

CONDITIONS: Advanced Unresectable Pancreatic Cancer
Keywords: Advanced; Unresesctable; Adenocarcinoma; Pancreatic cancer
MeSH Terms: conditions — Adenocarcinoma; Pancreatic Neoplasms | interventions — GV1001 peptide; Gemcitabine; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gemcitabine (Active Comparator): Gemcitabine alone treatment.
  Interventions: Drug: Gemcitabine (Chemotherapy)
- GV1001 (Experimental): GV1001 in sequential combination with Gemcitabine
  Interventions: Biological: GV1001

INTERVENTIONS:
Biological: GV1001 — 0.56mg GV1001 day 1, 3, 5, 8, 15, 22, week 6 and every 4 weeks thereafter. When gemcitabine is add it is given in cycles of once a week for 3 weeks and 1 week. Gemcitabine is dosed as per the SmPC.
  Other Names: INN-name: Termotide
  Arms: GV1001
Drug: Gemcitabine (Chemotherapy) — Gemcitabine is given as per the Burris regime and the SmPC, i.e. 7 weeks, followed by cycles of 1 weeks rest and 3 weeks chemotherapy.
  Other Names: Gemzar
  Arms: Gemcitabine

SUMMARY:
To investigate the efficacy of GV1001 in sequential combination with gemcitabine in locally advanced and metastatic adenocarcinoma of the pancreas.

DETAILED DESCRIPTION:
The trial is a Phase III, multinational, multicentre, controlled, randomised open-label trial. It will involve 520 advanced pancreatic cancer patients. Patients will be randomly assigned to receive Gemcitabine alone or GV1001 plus GM-CSF followed by addition of Gemcitabine at the time of 1st progression of disease. The experimental treatment is given prior to the current standard treatment in 50% of the patients.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed, unresectable, locally advanced, or metastatic adenocarcinoma of the pancreas.
2. Adequate hematological parameters:

   Hemoglobin >/= 9.5 g/dL [SI units, 5.9 mmol/L] WBC >/= 3000/mm3 [SI units, >/= 3 x 109/L] Platelets >/= 100,000/mm3 [SI units, >/= 100 x 109/L]
3. Adequate baseline liver function:

   Total Bilirubin < 3x ULN and

   Without liver metastases:

   AST (SGOT) </= 2.5 x ULN ALT (SGPT) </= 2.5 x ULN

   With liver metastases:

   AST (SGOT) </= 5 x ULN ALT (SGPT) </= 5 x ULN
4. Serum creatinine </= 1.5 mg/dL [SI units, 132 µmol/L].
5. Performance status ECOG 0-1.
6. Male or female 18 - 75 years inclusive.
7. Minimum life expectancy of 3 months.
8. Written informed consent.

Exclusion Criteria:

1. Treatment with chemotherapy for pancreatic cancer.
2. Treatment with other investigational drugs within the last 4 weeks prior to inclusion
3. Immune-suppressive therapy <4 weeks prior to inclusion
4. Chronic corticosteroid use except for asthma inhalers / topical use
5. Radiotherapy within 8 weeks of randomisation.
6. Other prior malignancies except for adequately treated non-melanoma skin cancers (BCC, SCC) and carcinoma in situ of the cervix.
7. Known diagnosis of HIV (AIDS), Hepatitis B, C.
8. Known history of or co-existing autoimmune disease.
9. Known CNS metastases.
10. Clinically significant serious disease or organ system disease not currently controlled on present therapy.
11. Pregnancy or lactation.
12. Women of childbearing potential not using reliable and adequate contraceptive methods*
13. Known sensitivity to any components of vaccine, gemcitabine or GM-CSF.
14. Unable for any other reason to comply with the protocol (treatment or assessments).

    * Adequate contraceptive methods are defined as the use of oral, implanted, injectable, mechanical or barrier products for the prevention of pregnancy; or women who are practising abstinence; or where the partner is sterile, for example a vasectomy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2006-06; Primary Completion 2008-08 (Estimated); Study Completion 2008-08 (Estimated)

PRIMARY OUTCOMES:
Overall survival time | 12 month

SECONDARY OUTCOMES:
Progression Free Survival | Time of progression

CONTACTS AND LOCATIONS:
Overall Officials: Ask Aabenhus, MSc. (Pharm), Study Director — Pharmexa A/S
Locations (86):
- United States (19):
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Genesis Cancer Center, Hot Springs, Arkansas
  - Scripps Clinic Torrey Pines, La Jolla, California
  - Desert Hematology Oncology Medical Group, Inc., Rancho Mirage, California
  - The Center for Hematology-Oncology, Boca Raton, Florida
  - Tampa General Hospital Usf Digestive Disorders Centre, Tampa, Florida
  - Palm Beach Cancer Institute, West Palm Beach, Florida
  - Portneuf Cancer Center, Pocatello, Idaho
  - Oncology Hematology Associates of Central Illinois, PC, Peoria, Illinois
  - Hematology Oncology Specialists, Covington, Covington, Louisiana
  - Berskhire Hematology Oncology PC, Pittsfield, Massachusetts
  - Billings Clinic, Billings, Montana
  - Carolinas Hematology Oncology Associates, Charlotte, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - Southwest Regional Cancer Center, Austin, Texas
  - Mary Crowley Medical Research Center (MCMRC)Texas Oncology-Presbyrerian Hospital of Dallas, Dallas, Texas
  - Mary Crowley Medical Research Center, Worth St., Dallas, Texas
  - Oncology Consultants, PA, Houston, Texas
- Australia (13):
  - St George Hospital, Department of Medical Oncology, Kogarah, New South Wales
  - Westmead Hospital, Dept. of Medical Oncology and Palliative Care, Westmead, New South Wales
  - The Townsville Hospital, Townsville Cancer Centre, Douglas, Queensland
  - Flinders Medical Centre, Medical Oncology - Clinical Trials, Bedford Park, South Australia
  - Dept. of Clinical Haematology / Oncology,the Queen Elizabeth Hospital, Woodville South, South Australia
  - Royal Hobart Hospital, Centre for Clinical Research, Hobart, Tasmania
  - Box Hill Hospital, ECRU Oncology, Box Hill, Victoria
  - The Alfred Hospital, Medical Oncology Unit, Melbourne, Victoria
  - Fremantle Hospital, Haemtology Department, Fremantle, Western Australia
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - Mount Medical Centre, Perth Oncology, Perth, Western Australia
  - Royal Perth Hospital, Department of Medical Oncology, Perth, Western Australia
  - Wesley Research Institute Limited, Auchenflower QLD
- Belgium (3):
  - Erasms University Hospital, Brussels
  - Hospital De Jolimont, Brussels
  - Ghent University Hospital, Digestive Oncology, Ghent
- Denmark (3):
  - Oncology Department, Århus Hospital, Aarhus
  - Oncology Department, Herlev Hospital, Herlev
  - Odense Universitetshospital, Onkologisk afd. R, Odense
- France (10):
  - Centre d'Etudes Cliniques en Oncologie, Centre Paul Papin, Angers
  - Oncologie Medicale, Clinic Pasteur, Évreux
  - Hepatogastroenterology Dpt, University Hospital Center of Grenoble, Grenoble
  - Service de Medicine Interne, CHRU de Lille, Lille
  - Oncologie Midicale CHR Lorient, Lorient
  - Hôpital de la Roche / Yon <<Les Oudaires>>, Centre Hospitalier Départmentale, Moreau
  - Oncologie Médicale, Centre Cathrine de Siennes, Nantes
  - Service de Cancerologie, Hospital Europeen Georges Pompidou, Paris
  - Medical Oncology Dpt, Armoricaine Private Hospital of Radiology, Saint-Brieuc
  - Clinic Saint Vincent, Saint-Grégoire
- Ireland (5):
  - Oncology Trials Unit, Cork University Hospital, Cork
  - Cancer Clinical Trials Unit, Beaumont Hospital, Dublin
  - Cancer Research Unit, Mater Misericordlae University Hospital, Dublin
  - Department of Medical Oncology, Amnch, Dublin
  - Oncology Research Team, Mater Private University Hospital, Dublin
- Italy (5):
  - Medical Oncology, University "Politecnica Delle Marche", Oncologia Medica Universita, Ancona
  - Policlinico Universitario "Mater Domini", Unita Oncologia, Catanzaro
  - Hospital "Careggi", Medical Oncology, Florence
  - Azienda Ospedaliera, Arcispedale S. Maria Nuova, Reggio Emilia
  - Hospital "G.B. Rossi", Surgical and Gastroenterological Dept. Borgo Roma, Verona
- VU University Medical Center, Amsterdam, Netherlands
- Norway (4):
  - Department of Oncology, Haukeland University Hospital, G.I. & Urogenital Oncology, Bergen
  - Sorlandet Hospital, Senter for Kreftbehandling, Kristiansand
  - Ullevål Universitetssykehus, Gastrokirurgisk afd., Oslo
  - Department of Oncology, University Hospital of Northern-Norway, Tromsø
- Poland (7):
  - Bialstocki Osrodek Onkologiczny, Oddzial Chemioterapii Nowotworow I Chorob Wewnetrznych, Bialystok
  - W.S2.Z, Krolewiecka, Elblag
  - Wojewodzki Szpital Specjalistyczny im.Rydgiera, Oddzial Chemioterapii, Krakow
  - Klinika Chemioterapii Uniwersytetu Medycznego w Lodzi, Medical University, Lodz
  - Zaklad Opieki Zdrowotnej MSWiA, Olsztyn
  - Centrum Onkologii, Wosewodzki Osrodek Onkologii, Opole
  - Dolnoslaskie Centrum Onkologii, Oddzial Chemioterapii, Wroclaw
- Spain (11):
  - Hospital Clinic I Provincial De Barcelona, Barcelona
  - Medical Oncology Department, General Hospital of Baza, Granada
  - Medical Oncology Department, Virgen de Las Nieves Hospital, Granada
  - Hospital Universitario Gregorio Marañón, Departamento de Oncología, Madrid
  - Clínica Puerta de Hierro, Departamento de Oncología, Madrid
  - Hospital Universitario La Paz, Departamento de Oncología, Madrid
  - H. Monteprincipe, Madrid
  - Fundaciόn Hospital de Alcorcόn, Unidad de Oncología, Madrid
  - HRU Carlos Haya, Medical Oncology Unit, Málaga
  - Oncology Department, Clinic Universitary Hospital, Málaga
  - Digestive Unit, Universitary Hospital Virgen de La Macarena, Seville
- Sweden (5):
  - Sahlgrenska Hospital, Head Division for Upper GI Surgery, Gothenburg
  - University Hospital, Department Of surgery and Gasterenterology, Lund
  - Department of Oncology, Malmö University Hospital, Malmo
  - Karolinska Institute / Hospital Solna, Department of Oncology, Stockholm
  - Department of Oncology, Karolinska Universitetssjukhuset, Stockholm